CLINICAL TRIAL: NCT01500564
Title: Functional Interest of Non Invasive Brain Stimulation During Physiotherapy at a Subacute Phase Post Stroke (Anodal Protocol).
Brief Title: Functional Interest of Non Invasive Brain Stimulation During Physiotherapy at a Subacute Phase Post Stroke (Anodal Protocol): ReSTIM
Acronym: ReSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010.635
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Stroke
Keywords: Stroke; transcranial direct current stimulation (tDCS); motor function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham tDCS and motor training: sham comparator (Sham Comparator): Participants will receive sham tDCS over the primary motor cortex of the ipsilesional hemisphere during 20 minutes of motor training (10 consecutive sessions Monday-Friday during two weeks).
  Intervention: placebo tDCS Other: Motor Training
  Interventions: Device: Sham tDCS
- Anodal tDCS and motor training: experimental (Experimental): Participants will receive anodal tDCS over the primary motor cortex of the ipsilesional hemisphere. The following parameters will be used: stimulation intensity of 1mA during 20 minutes of motor training (10 consecutive sessions Monday-Friday during two weeks).
  Interventions:
  * Device: anodal tDCS
  * Other: motor Training during physiotherapy
  Interventions: Device: anodal tDCS (device) Eldith DC-Stimulator

INTERVENTIONS:
Device: anodal tDCS (device) Eldith DC-Stimulator — tDCS applied to the motor cortex every day of two consecutive weeks (10 sessions) at 1 mA during 20 minutes. Conductive rubber covered by sponges soaked in saline will be used, held in place by a band. The current will be gradually increased over 100 seconds.
  Other Names: Eldith DC-Stimulator (CE certified)
  Arms: Anodal tDCS and motor training: experimental
Device: Sham tDCS — Participants will receive sham tDCS over the primary motor cortex of the ipsilesional hemisphere during 20 minutes of motor training (10 consecutive sessions Monday-Friday during two weeks).
  Arms: Sham tDCS and motor training: sham comparator

SUMMARY:
Previous research that utilises single sessions of transcranial direct current stimulation (tDCS) have demonstrated functional improvements. However these improvements are usually short-lived, lasting less than one hour before the patient's performance returns to baseline. In these studies, tDCS is typically applied with the goal of adaptively enhancing functional activation of pathologically under-active tissue or suppressing pathologically over-active tissue. Interestingly, a small body of evidence is now emerging to indicate that tDCS can improve learning/memory functions in healthy controls. The goal of this study is to test if the application of tDCS could enhance learning and/or memory for physiotherapy rehabilitation, which may in turn lead to correspondingly greater motor improvement. Patients at a subacute stage (1 to 6 month post stroke) will attend for 10 consecutive daily sessions of tDCS.

This research has important implications; previous studies suggest that such an approach has the potential to facilitate physical rehabilitation post-stroke and establish tDCS as a clinically viable rehabilitative tool. Recovery of motor skills may take many months to acquire and therefore strategies that have the potential to enhance acquisition of skill are of practical and scientific interest.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be between the ages of 18-90 and must not be pregnant.
* Patients volunteer to participate in the study, with a written informed consent signed
* Affiliation to a national health insurance program
* First-time clinical ischemic or hemorrhagic cerebrovascular accident - evidenced by a radiological (or physician's) report
* Contralesional motor deficit
* Lesion sparing primary motor cortex
* Stroke onset >1 month and <6 months prior to study enrollment

Exclusion Criteria:

* Coexistent major neurological or psychiatric disease as to decrease number of confounders
* History of epilepsy before stroke (or episodes of seizures within the last six months)
* Any substantial decrease in alertness, language reception, or attention that might interfere with understanding instructions for motor testing
* Subjects with global aphasia and deficits of comprehension
* Excessive pain in any joint of the paretic extremity (VAS>4)
* Contraindications to Tdcs : metal in the head, implanted brain medical devices
* Coexistent major neurological or psychiatric disease as to decrease number of confounders
* A history of significant alcohol or drug abuse in the prior 6 months
* Anyone who is currently taking or who has taken anti-malarial treatment in the last 72 hours
* Subjects may not have already received constraint induced motor therapy and/or tDCS treatment for stroke
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01-02 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment (Upper extremity) of motor recovery following stroke | assessed at one baseline session (day 4), and then again immediately following the last day of the intervention (day 18), 2 weeks (day 32), 1 month, 3 months and 6 months later.
  Main primary outcome is change in score between the baseline session score and day 32.

SECONDARY OUTCOMES:
Functional independence scale (MIF) | assessed at one baseline session (day 4), and then again immediately following the last day of the intervention (day 18), 2 weeks (day 32), 1 month, 3 months and 6 months later.
  We are looking for a change in scores between the baseline session score, and those collected during each follow-up session.
Motor Activity Log (MAL) | assessed at one baseline session (day 4), and then again immediately following the last day of the intervention (day 18), 2 weeks (day 32), 1 month, 3 months and 6 months later.
  We are looking for a change in scores between the baseline session score, and those collected during each follow-up session.
Jebsen Taylor Hand function test (JTT) | assessed at one baseline session (day 4), and then again immediately following the last day of the intervention (day 18), 2 weeks (day 32), 1 month, 3 months and 6 months later.
  We are looking for a change in scores between the baseline session score, and those collected during each follow-up session.
Box and block test (BBT) | assessed at one baseline session (day 4), and then again immediately following the last day of the intervention (day 18), 2 weeks (day 32), 1 month, 3 months and 6 months later.
  We are looking for a change in scores between the baseline session score, and those collected during each follow-up session.
Modified Ashworth Scale | assessed at one baseline session (day 4), and then again immediately following the last day of the intervention (day 18), 2 weeks (day 32), 1 month, 3 months and 6 months later.
  We are looking for a change in scores between the baseline session score, and those collected during each follow-up session.
Testing motor MRC | assessed at one baseline session (day 4), and then again immediately following the last day of the intervention (day 18), 2 weeks (day 32), 1 month, 3 months and 6 months later.
  We are looking for a change in scores between the baseline session score, and those collected during each follow-up session.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie JACQUIN-COURTOIS, MD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Centre de Lay-Saint-Christophe-Institut Régional de Médecine Physique et de Réadaptation, Lay-Saint-Christophe
  - Hospices Civils de Lyon- Hôpital Henry Gabrielle-Service de Médecine Physique et Réadaptation, Saint-Genis-Laval

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411